CLINICAL TRIAL: NCT02971748
Title: A Phase II Study of Anti-PD-1 (Pembrolizumab) in Combination With Hormonal Therapy During or After Radiation in Patients With Hormone Receptor (HR)-Positive Localized Inflammatory Breast Cancer (IBC) Who Did Not Achieve a Pathological Complete Response (pCR) to Neoadjuvant Chemotherapy
Brief Title: Pembrolizumab in Treating Patients With Hormone Receptor Positive, Localized Inflammatory Breast Cancer Who Are Receiving Hormone Therapy and Did Not Achieve a Pathological Complete Response to Chemotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0096; NCI-2018-01297 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0096 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Breast Inflammatory Carcinoma; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: conditions — Inflammatory Breast Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab works in treating patients with hormone receptor positive inflammatory breast cancer that has not spread to other parts of the body, who are receiving hormone therapy and did not achieve a pathological complete response to chemotherapy. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the disease free survival (DFS) at 2 years of patients with maintenance therapy using pembrolizumab in combination with standard adjuvant hormonal therapy.

II. To determine the safety and toxicity profile of primary inflammatory breast cancer (IBC) patients who received combination of pembrolizumab and hormone receptor blockade.

EXPLORATORY OBJECTIVES:

I. To investigate the association between immune related biomarkers in the peripheral blood and tumor tissue, such as PD-L1 expression, with safety and efficacy for IBC patients treated with pembrolizumab.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Is willing and able to provide written informed consent for the trial.
2. Is a female or male and >/= 18 years of age
3. Has histological confirmation of breast carcinoma.
4. Has confirmed inflammatory breast cancer by using international consensus criteria:

   * Onset: Rapid onset of breast erythema, edema and/or peau d'orange, and/or warm breast, with/without an underlying breast mass
   * Duration: History of such findings no more than 6 months
   * Extent: Erythema occupying at least 1/3 of whole breast
   * Pathology: Pathologic confirmation of invasive carcinoma
5. Did not achieve pathological complete response (pCR) to any chemotherapy that was given with the intention to induce best response prior surgery. pCR is defined as the current American Joint Committee on Cancer (AJCC) breast cancer staging.
6. Is HER2 normal, defined as HER2 0 or 1+ by IHC and negative by FISH if performed; or HER2 is 2+ by IHC and negative by FISH; or HER2 negative by FISH if IHC is not performed.
7. Has positive ER or PR status. ER or PR >/= 10%
8. Has a performance status of 0-1 on the ECOG Performance Scale.
9. Has adequate organ function as determined by the following laboratory values:

   ANC >/= 1,500 /mcL, Platelets >/=100,000 /mcL, Hgb >/= 9 g/dL, creatinine levels < 1.5 x ULN, Total bilirubin </= 1.5 x ULN, ALT and AST </= 2.5 x ULN
10. Participants of reproductive potential must agree to avoid becoming pregnant or impregnating a partner, respectively, while receiving study drug and for 120 days after the last dose of study drug by complying with one of the following: (1) practice abstinence† from heterosexual activity; OR (2) use (or have their partner use) acceptable contraception during heterosexual activity.

Acceptable methods of contraception are: Single method (one of the following is acceptable): (1) intrauterine device (IUD); (2) vasectomy of a female participant's male partner; (3) contraceptive rod implanted into the skin. Combination method (requires use of two of the following): (1) diaphragm with spermicide (cannot be used in conjunction with cervical cap/spermicide); (2) cervical cap with spermicide (nulliparous women only); (3) contraceptive sponge (nulliparous women only); (4) male condom or female condom (cannot be used together); (5) hormonal contraceptive: oral contraceptive pill (estrogen/progestin pill or progestin-only pill), contraceptive skin patch, vaginal contraceptive ring, or subcutaneous contraceptive injection.

Female participants will be considered of non-reproductive potential if they are either:

(1) postmenopausal (defined as at least 12 months with no menses without an alternative medical cause; in women < 45 years of age a high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. In the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.); OR (2) have had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy or bilateral tubal ligation/occlusion, at least 6 weeks prior to screening; OR (3) has a congenital or acquired condition that prevents childbearing.

Male participants will be considered to be of non-reproductive potential if they have azoospermia (whether due to having had a vasectomy or due to an underlying medical condition).

11. Has negative serum or urine pregnancy test for subjects of childbearing potential within 10 days before first dose.

12. Have completed radiation (if candidate for post-mastectomy radiation) or plans to begin radiation and endocrine therapy within 28 days.

13. If the participant has already started hormonal blockade therapy after radiation as adjuvant therapy, the patient is eligible as long as the hormonal therapy was initiated no more than 6 months before the screening day and the participant can start the study drug within 4 weeks since the completion of screening.

Exclusion Criteria:

1. Is currently participating in a study of an investigational anti-cancer agent.
2. Has a diagnosis of immunodeficiency or any other form of immunosuppressive therapy.
3. Has not recovered from adverse events due to prior therapies, i.e. monoclonal antibody, chemotherapy, targeted small molecule therapy, radiation therapy, or surgery.

   - Note: Participants with ≤ Grade 2 neuropathy, alopecia and general disorders and administration site conditions (per CTCAE version 4.0) are an exception to this criterion and may qualify for the study.
4. Has a known history of prior malignancy with the exception of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, or in situ cervical cancer, and has undergone potentially curative therapy and has no evidence of recurrence over the last 1 year since completion of curative therapy.
5. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or immunosuppressive agents. Participants with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Participants that require intermittent use of bronchodilators, inhaled steroid or local steroid injections to the skin would not be excluded from the study. Participants with hypothyroidism stable on hormone replacement or Sjögren's syndrome will not be excluded from the study.
6. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
7. Has an active infection requiring systemic therapy.
8. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
9. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
10. Has a known history of Human Immunodeficiency Virus (HIV).
11. Has a known active Hepatitis B or Hepatitis C
12. Have received a live vaccine within 30 days prior to the first dose of trial treatment.
13. Gastrointestinal tract disease or defect or previous history of colitis.
14. Has proven or suspected distant metastasis that involves occurrence of breast cancer outside of loco-regional breast and lymph nodes area.
15. Participants requiring daily corticosteroids either via po or infusion
16. Myocardial infarction within 6 months before starting therapy, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or unstable cardiac arrhythmia requiring medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2027-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bora Lim, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Mar 2017~ Sept 2025. All recruitment was done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: 36 patients were accrued and assessed for eligibility and 31 patients were assigned to the cohort.
Groups:
- Pembrolizumab + Hormonal Therapy for HR+ Localized IBC Without pCR After Neoadjuvant Chemo: Pembrolizumab 200 mg every 3 weeks with hormonal therapy per physician discretion.
Period: Overall Study
Arm/Group | Pembrolizumab + Hormonal Therapy for HR+ Localized IBC Without pCR After Neoadjuvant Chemo
Started | 31
Completed | 8
Not Completed | 23
Not completed — Adverse Event | 12
Not completed — Withdrawal by Subject | 1
Not completed — Financial issue | 2
Not completed — Clinical progression | 8

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab + Hormonal Therapy for HR+ Localized IBC Without pCR After Neoadjuvant Chemo
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 25
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS)
Description: Disease-free survival (DFS) is defined as the time from treatment initiation to recurrence of disease or death from any cause. Patients without an event were censored at their last disease assessment.
Time Frame: From treatment initiation through last available follow-up (up to approximately 9 years)
Population: All treated patients were included in the DFS analysis.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Pembrolizumab + Hormonal Therapy for HR+ Localized IBC Without pCR After Neoadjuvant Chemo
Number analyzed (Participants) | 31
years | 4.22 [2.17 to NA] — The upper confidence limit was not estimable because insufficient progression events occurred after the median time point.

2. Primary Outcome: Participants With Treatment-Related Adverse Events
Description: Number of participants experiencing treatment-related adverse events, graded according to CTCAE v4.0.
Time Frame: From first dose through 30 days after last dose (up to approximately 25 months)
Population: All treated patients were included in the safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Hormonal Therapy for HR+ Localized IBC Without pCR After Neoadjuvant Chemo
Number analyzed (Participants) | 31
Participants
  Abdominal pain | 1
  Alanine aminotransferase increased | 1
  Anorexia | 1
  Arthralgia | 7
  Aspartate aminotransferase increased | 1
  Colitis | 4
  Cough | 2
  Diarrhea | 3
  Dry mouth | 1
  Dyspnea | 1
  Esophagitis | 1
  Fatigue | 7
  Hyperglycemia | 1
  Hyperkalemia | 1
  Hypertriglyceridemia | 1
  Hypothyroidism | 9
  Positive ANA antibody | 1
  Joint effusion | 1
  Lymphocyte count decreased | 2
  Myalgia | 2
  Nausea | 3
  Osteoporosis | 1
  Palmar-plantar erythrodysesthesia syndrome | 1
  Pneumonitis | 4
  Pruritus | 2
  Rash maculo-papular | 3
  Urinary tract infection | 1

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed for up to 2 years after treatment discontinuation. Adverse events were assessed from first protocol-specific intervention through 30 days after last pembrolizumab dose (up to approximately 25 months)
Description: Adverse events were assessed using CTCAE v4.0. All AEs of ≥ Grade 2 for non-hematologic events and ≥ Grade 3 for hematologic events, regardless of attribution, were recorded.
Arm/Group | Pembrolizumab + Hormonal Therapy for HR+ Localized IBC Without pCR After Neoadjuvant Chemo
All-Cause Mortality (participants affected / at risk) | 9/31
Serious Adverse Events (participants affected / at risk) | 6/31
Other Adverse Events (participants affected / at risk) | 28/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab + Hormonal Therapy for HR+ Localized IBC Without pCR After Neoadjuvant Chemo (N=31)
Colitis (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab + Hormonal Therapy for HR+ Localized IBC Without pCR After Neoadjuvant Chemo (N=31)
Hypothyroidism (Endocrine disorders) | 9
Eye pain (Eye disorders) | 1
Retinal vascular disorder (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Bloating (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Oral pain (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 9
Flu like symptoms (General disorders) | 2
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 2
Positive ANA antibody (Immune system disorders) | 1
Bladder infection (Infections and infestations) | 1
Bronchial infection (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
COVID-19 infection (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 4
Tooth infection (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
INR increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 3
Weight gain (Investigations) | 1
Weight loss (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 11
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hip pain (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2
Cognitive disturbance (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Balance difficulty (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 9
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT02971748/Prot_SAP_000.pdf